



This letter serves to confirm that the study protocol entitled "Marginal Bone Loss Around Bone-Level & Tissue-Level Dental Implants" under the direction of Principal Investigator Ahmed Samir Mabrouk Oraby Elkattan, has been reviewed and granted full approval by the Comitè d'Ètica i Investigació amb Medicaments de l'Hospital Odontològic Universitat de Barcelona (CEIm HOUB).

The approval was granted on September 28, 2022, under the official approval number 33-2022.

The associated informed consent form, dated July 1, 2022, was reviewed and approved by this committee as part of the protocol evaluation.

This document is attached for your records.

Please do not hesitate to contact us at ceic.hospitalodontologic@ub.edu if you require any further information or verification.

Sincerely,

LOPEZ Firmado digitalmente por LOPEZ LOPEZ JOSE - 40962929K Fecha: 2025.07.21 18:01:52 +02'00'

Atentamente,

José López López Profesor Titular de Medicina Oral Director facultativo del Hospital Odontológico Universidad de Barclona Universidad de Barcelona Comitè d'Ètica i Investigació amb Medicaments (CEIm HOUB)

ceic.hospitalodontologic@ub.edu

+34 606 457 362





## **CONSENTIMENT INFORMAT PARTICIPANT ESTUDI**

| Study title:<br>MARGINAL BONE LOSS: IMPLAN | ITS AT TISSUE LEVEL AND E | BONE LEVEL |
|---|---|---|
| | representative, family me | mber, etc. of the participant, the |
| I <b>DECLARE</b> that Dr. AHMED SAMIR MABROUK ORABY ELKATTAN (Name and two surnames of the researcher who provides the information) You have provided sufficient information about the study and that has been submitted to the corresponding Full of Information. | | |
| Here are the explanations that have been provided to me in a clear and user-friendly language, and the faculty member has allowed me to make all of the observations and has clarified all of the doubts that I have raised. | | |
| I also understand that, at any time when I feel the need to donate explanations, I can revoke the consent that has been granted and can withdraw from the study as I speak, without having to donate explanations and without any repercussions. | | |
| For this reason, I declare that I am satisfied with the information provided and that I give my consent to participate in this study. | | |
| Signature<br>Investigator | Signature<br>Participant | Signature<br>Legal Representative Participant |
| L'Hospitalet de Llobregat, of of 20 | | |







## **CONSENTIMENT INFORMAT PARTICIPANT ESTUDI**

| REVOCATION OF CONSENT | | |
|---|---|---|
| Mr./Mrs | | as a participant |
| with DNI | or as legal representative, family, etc. of the participant, | |
| Mr./Mrs | with DNI no | |
| I DECLARE that: | | |
| The Dr | | |
| You have informed me correctly about the study | | |
| I REVOCATE consent | | |
| L'Hospitalet de Llobregat, de de 20 | | |
| Signature | Signature | Signature |
| Reasearcher | Participant | Participating Legal representative |

